CLINICAL TRIAL: NCT02210702
Title: Oral Contraceptive Ethinyl Estradiol Dose Effect on Postpartum Depression and Sexual Functioning Scales
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Jones Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 14-06-FB-0118-HOSP
Record Dates: First submitted 2014-07-31; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Postpartum Depressive Mood; Postpartum Sexual Function
MeSH Terms: interventions — Ethinyl Estradiol; Norethindrone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ethinyl Estradiol 35mcg/Noethindrone 1mg (Experimental): 21 day supply of Ethinyl Estradiol 35mcg/Norethindrone 1mg will be taken beginning at Week 3 postpartum
  Interventions: Drug: Ethinyl Estradiol 35mcg/Norethindrone 1mg
- Ethinyl Estradiol 20mcg/Norethindrone 1mg (Experimental): 21 day supply of Ethinyl Estradiol 20mcg/Norethindrone 1mg will be taken beginning at Week 3 postpartum
  Interventions: Drug: Ethinyl Estradiol 20mcg/Norethindrone 1mg
- No hormonal contraception (No Intervention): Women choosing copper IUD, spermicides, barrier methods, or sterilization (tubal ligation or partner vasectomy).

INTERVENTIONS:
Drug: Ethinyl Estradiol 35mcg/Norethindrone 1mg
  Arms: Ethinyl Estradiol 35mcg/Noethindrone 1mg
Drug: Ethinyl Estradiol 20mcg/Norethindrone 1mg
  Arms: Ethinyl Estradiol 20mcg/Norethindrone 1mg

SUMMARY:
This is a prospective, randomized, controlled cohort study. This study will look at the effect of Ethinyl Estradiol 35mcg/Norethindrone 1mg and Ethinyl Estradiol 20 mcg/Norethindrone 1mg on postpartum depressive symptoms and sexual function scores when compared to a control group using no hormonal contraception. Depressive symptoms and sexual function will be measured using the Edinburgh Postnatal Depression Scale (EPDS), Arizona Sexual Experiences Scale (ASEX), and Brief Index of Sexual Functioning for Women (BISF-W). Participants will begin taking the medication at Week 3 postpartum, and these outcomes will be measured at baseline (0-1 day postpartum), Week 3, and Week 6-7. The investigators hypothesize that there will be an ethinyl estradiol dose related response in EPDS, ASEX, and BISF-W scores at Week 6-7, which would indicate a decrease in depressive symptoms and increase in sexual function in both of the oral contraceptive groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 year old women who desire contraception postpartum for at least 6 weeks.
* 18-45 year old women who choose not to use oral contraceptive medication postpartum for at least 6 weeks for the control group.

Exclusion Criteria (Medication groups):

* Breastfeeding (although this may limit participant enrollment, combined oral contraceptives are contraindicated in this population).
* Delivery by cesarean section.
* Previous history of depression, mood disorders, or psychiatric disorders.
* Any condition (history or presence of) which contraindicates the use of combination OCs, including:
* Thrombophlebitis or thromboembolic disorders, known or suspected clotting disorders, deep vein thrombosis, thrombogenic valvulopathies or rhythm disorders.
* Pulmonary Embolism.
* Cerebrovascular or coronary artery disease or myocardial infarction.
* Diabetes mellitus.
* Migraine headaches with focal, neurological symptoms.
* Chronic renal disease.
* Uncontrolled or untreated hypertension.
* Cholestatic jaundice.
* Known or suspected carcinoma of the breast, endometrial carcinoma, or known or suspected estrogen-dependent neoplasia.
* Impaired liver function or disease, hepatic adenomas or carcinomas.
* Known hypersensitivity to estrogens and/or progestins.
* History of thyroid disorders.
* Recent alcohol or drug use.
* Smoking and age ≥35 or smokers who will become 35 years of age during the study.
* Known history of noncompliance with taking medication.

Exclusion Criteria (Control group):

* Previous history of depression, mood disorders, or psychiatric disorders.
* Recent alcohol or drug use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Change in Edinburgh Postnatal Depression Scale at baseline, 3 weeks postpartum and 6 weeks pospartum | Baseline (0-1 days postpartum), Week 3 Postpartum, Week 6-7 Postpartum
Change in Arizona Sexual Experiences Scale scores at baseline, 3 weeks postpartum, and 6-7 weeks postpartum | Baseline (0-1 days postpartum), Week 3 Postpartum, Week 6-7 Postpartum
Change in Brief Index of Sexual Functioning for Women scores at baseline, week 3 postpartum, and week 6-7 postpartum | Baseline (0-1 days postpartum), Week 3 Postpartum, Week 6-7 Postpartum

SECONDARY OUTCOMES:
Time to First Coitus | Time to first coitus during postpartum period
Urine Pregnancy Test | Week 6-7 Postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States